CLINICAL TRIAL: NCT04860154
Title: Evaluation of Bile Duct Patency After Photodynamic Therapy in Unresectable Cholangiocarcinoma：a Prospective Non-randomized Controlled Study
Brief Title: Photodynamic Therapy for Cholangiocarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Principal Investigator, Xun Li, Director，M.D., Ph.D., Hepatopancreatobiliary Surgery Institute of Gansu Province
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Photodynamic therapy
Record Dates: First submitted 2021-04-17; First posted 2021-04-26 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Cholangiocarcinoma Non-resectable
Keywords: ERCP; PDT; Cholangiocarcinoma; Bile duct drainage; Stent
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Hematoporphyrins

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PDT with stent (Experimental): Before photodynamic therapy, candidate patients undergoing biliary biopsy and biliary duct drainage. If pathology shows a bile duct malignancy, PDT therapy will carry out until total bilirubin drops below 100 μmol/L.Patients with negative skin test of hematoporphyrin Injection (3.0-5.0mg/Kg plus saline 250 mL intravenous drip, the drip was completed within 1 hour) and keep patients away from the light. The first PDT therapy was performed 24 hours after infusion of hematoporphyrin injection by ERCP. The biliary tumor necrosis was observed and the biliary tract was cleaned up 24 hours later and then PDT therapy showed again if necessary. Multiple plastic stents or metal stent will be placed. Follow up regularly after the procedure, PDT therapy would be given again in 3 months.
  Interventions: Drug: Hematoporphyrin
- ERCP stent (No Intervention): After obtaining bile duct biopsy, the candidates were placed with biliary plastic stents or metal stents directly.

INTERVENTIONS:
Drug: Hematoporphyrin — Patients with negative skin test of hematoporphyrin Injection (3.0-5.0mg/Kg plus saline 250 mL intravenous drip, the drip was completed within 1 hour) and keep patients away from the light. The first PDT therapy was performed 24 hours after infusion of hematoporphyrin injection by ERCP. The biliary tumor necrosis was observed and the biliary tract was cleaned up 24 hours later and then PDT therapy showed again if necessary. Multiple plastic stents or bald metal stents will be placed. Follow up regularly after the procedure, PDT therapy would be given again in 3 months.
  Other Names: ERCP stents
  Arms: PDT with stent

SUMMARY:
Comparison of the bile duct patency with photodynamic therapy (PDT) and regular Endoscopic Retrograde Cholangiopancreatography(ERCP) stents in unresectable cholangiocarcinoma.

DETAILED DESCRIPTION:
Cholangiocarcinoma is a malignant tumor originating from the bile duct epithelium, accounting for about 70% of the malignant tumors of the bile duct system. Patients have no obvious clinical symptoms in the early stage. After late diagnosis, the effective treatment is surgical resection and & or liver transplantation, and chemotherapy is only used as adjuvant or palliative treatment. Some types of cholangiocarcinomas, such as hilar cholangiocarcinomas, are difficult to achieve radical resection due to their anatomical location, early invasions and are prone to recurrence with a poor long-term efficacy after surgery. Therefore, the comprehensive treatment of cholangiocarcinoma by multiple means urgently needs to be explored. In recent years, photodynamic therapy (PDT), as a new local treatment method, has attracted increasing attention.

This study investigates the bile duct patency and effectiveness of photodynamic therapy compare with ordinary ERCP treatment for cholangiocarcinoma including the median survival, overall survival, and other indicators of side effects.

ELIGIBILITY:
Inclusion Criteria:

* ERCP cholangiocarcinoma（the tumor is unresectable or patient can't accept surgery in the situation, the tumor can be resected but the patients cannot tolerate surgery）;

Exclusion Criteria:

* Proximal cholangiocarcinoma (Bismuth type Ⅲ-Ⅳ, or intra-hepatic cholangiocarcinoma);
* Patients with Karnofsky Performance Scale (KPS) score≤70；
* Expected survival≤3months；
* Patients with porphyria；
* Coagulation dysfunction (INR> 1.5) and low peripheral blood platelet count(<50×10^9 / L) or using anti-coagulation drugs；
* Bilirubin could not be reduced to less than 100mmol/L within 1 month after drainage；
* Patients have intrahepatic metastasis or distant metastasis；
* Patients with no pathological diagnosis；
* known to allergic to study drug(porphyrin drugs) or other similar and related compounds；
* Other photosensitizers have been used within 4 weeks prior；
* Metal biliary stents were placed previously；
* Patients with contraindications to ERCP；
* Patients with HIV infection；
* Pregnant, parturient, or breastfeeding women；
* Patients complicated with other malignant tumors；
* Patients with severe liver function damage；
* Patients who were in cachexia, liver abscess, or advanced patients who were unable to tolerate PDT；
* Patients with other serious physical or mental illnesses that prevent researchers to enroll them in this study as subjects；
* Patients with other contraindications for photodynamic therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2021-04-17 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Bile duct patency | 3years (every 3 months or obstruction appears)
  Patency period of the stents after treatment
Median survival time | 3years (every 3 months）
  The time of the half of the patients survived after initial therapy

SECONDARY OUTCOMES:
Overall survival | 5years (every 3 months）
  The time from initial therapy to death or the end of the study
Karnofsky Performance Scale | 1year (baseline and every 3 months）
  The Karnofsky Performance Scale scores range from 0 (death) to 100 (normal). The lower the Karnofsky score, the worse likelihood of survival. However, the premature termination of the study does not allow for a meaningful analysis of the scale where 100% means no complaints with no evidence of disease, 80% is a normal activity with effort and some signs or symptoms of the disease. pre-operation, 1 month, 3 months, 6 months, 9 months, and 12 months after the operation
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 | 1year (baseline and every 3 months）
  EORTCQLQ-C30 score used to assess the quality of life of cancer patients. EORTCQLQ-C30 score contains 30 questions, the first 28 questions include 1-4 points, the lower the score, the better; but the latter two questions include 1-7 points, the higher the score, the better. pre-operation, 1 month, 3 months, 6 months, 9 months, and 12 months after the operation
The change of weight in kilograms | 1year (baseline and every 3 months）
  Weight changes of the patient before and after PDT treatment, pre-operation, 1 month, 3 months, 6 months, 9 months, and 12 months after the operation
Beck Anxiety Inventory | 1year (baseline and every 3 months）
  BAI is a 21-item self-reported questionnaire that measures the existence and severity of symptoms of anxiety. Each of the 21 items on the BAI tool represents an anxiety symptom. A total score of 0 - 7 is interpreted as a "Minimal" level of anxiety; 8 - 15 as "Mild"; 16 - 25 as "Moderate", and; 26 - 63 as "Severe", pre-operation, 1 month, 3 months, 6 months, 9 months and 12 months after the operation
Cumulative treatment costs | 5years (baseline and in each year）
  The overall treatment costs from initial PDT to death or the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Xun Li, M.D.,Ph.D., Study Chair — Hepatopancreatobiliary Surgery Institute of Gansu Province
Locations (11):
- China (11):
  - Southwest Hospital, Army Medical University, Chongqing, Chongqing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Hospital of Jilin University, Changchun, Jilin
  - General Hospital of Ningxia Medical University, Yingchuan, Ningxia
  - The first affiliated hospital of Xi 'an JiaoTong university, Xi'an, Shaanxi
  - Shandong Provincial Third Hospital, Jinan, Shandong
  - Xinhua Hospital, Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - General Hospital of Taiyuan Iron and Steel Corporation, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu Y, Liu L, Wu JC, Bie LK, Gong B. Efficacy and safety of photodynamic therapy for unresectable cholangiocarcinoma: A meta-analysis. Clin Res Hepatol Gastroenterol. 2015 Dec;39(6):718-24. doi: 10.1016/j.clinre.2014.10.015. Epub 2015 Jun 10. PMID 26070572
- [Background] Gonzalez-Carmona MA, Bolch M, Jansen C, Vogt A, Sampels M, Mohr RU, van Beekum K, Mahn R, Praktiknjo M, Nattermann J, Trebicka J, Branchi V, Matthaei H, Manekeller S, Kalff JC, Strassburg CP, Weismuller TJ. Combined photodynamic therapy with systemic chemotherapy for unresectable cholangiocarcinoma. Aliment Pharmacol Ther. 2019 Feb;49(4):437-447. doi: 10.1111/apt.15050. Epub 2019 Jan 13. PMID 30637783
- [Background] Strand DS, Cosgrove ND, Patrie JT, Cox DG, Bauer TW, Adams RB, Mann JA, Sauer BG, Shami VM, Wang AY. ERCP-directed radiofrequency ablation and photodynamic therapy are associated with comparable survival in the treatment of unresectable cholangiocarcinoma. Gastrointest Endosc. 2014 Nov;80(5):794-804. doi: 10.1016/j.gie.2014.02.1030. Epub 2014 May 15. PMID 24836747
- [Background] Talreja JP, Degaetani M, Ellen K, Schmitt T, Gaidhane M, Kahaleh M. Photodynamic therapy in unresectable cholangiocarcinoma: not for the uncommitted. Clin Endosc. 2013 Jul;46(4):390-4. doi: 10.5946/ce.2013.46.4.390. Epub 2013 Jul 31. PMID 23964337